CLINICAL TRIAL: NCT00163800
Title: Outcome Predictors in Acute Brain Injury, A Pilot Study
Brief Title: Outcome Predictors in Acute Brain Injury
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Other Study IDs: 189/02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-12-08 (Estimated); Status verified 2005-09

CONDITIONS: Acute Brain Injury
Keywords: Outcome predictors; Acute brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study will attempt to evaluate clinical, laboratory and radiographic parameters together to assess heir values in outcome prediction from brain injury. Patients will be followed up for a period of 6 months, following admission to ICU, to assess outcome, using the Extended Glasgow Outcome Score (GOSE).

We hypothesise that it is possible to reliably predict outcome in brain injury from the current investigations we have at our disposal.

DETAILED DESCRIPTION:
Design- A prospective clinical trial of patients admitted to intensive care with acute brain injury due to trauma.

Setting- Intensive Care Unit of the Alfred Hospital Clinical Examination- Day 4 and day 8, ICU consultant to assess prognosis and score patient.

Electrophysiology- Day 4 and day 8, SSEP and EEG. Interpretation by person blinded to the patient.

CT Brain- Day 1, day 4 and day 8. Interpretation by radiologist blinded to the patient.

Blinding- Persons blinded to the patients will make all interpretations of investigations. Mode of brain injury will be made available.

Follow up of patients- Structured interviews by telephone will be performed at 6 months post injury with the patient alone, relatives/ friend/ carer alone or patient and relatives/ friend/ carer. These will be performed in relation to the Extended Glasgow Outcome Scale (GOSE).

Statistics- The positive and negative predictive values for the tests will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale < 9 post resuscitation
* Intubated and ventilated
* Traumatic brain injury

Exclusion Criteria:

* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-07; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Warwick Butt, FRACP, Principal Investigator — Bayside Health